CLINICAL TRIAL: NCT03837184
Title: Phase 3, Open-Label, Single-Arm, Single-Dose Gene Replacement Therapy Clinical Trial for Patients With Spinal Muscular Atrophy Type 1 With One or Two SMN2 Copies Delivering AVXS-101 by Intravenous Infusion
Brief Title: Single-Dose Gene Replacement Therapy Using for Patients With Spinal Muscular Atrophy Type 1 With One or Two SMN2 Copies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Gene Therapies (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVXS-101-CL-306; 194664 (Other: JapicCTI); 201900208 (Other: Ministry of Food and Drug Safety (South Korea)); COAV101A12304 (Other: Novartis Pharmaceuticals)
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Results first posted 2022-01-11 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Spinal Muscular Atrophy Type I
Keywords: Spinal Muscular Atrophy; SMN2; Onasemnogene Abeparvovec-xioi; Gene replacement therapy
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood; Muscular Atrophy, Spinal | interventions — Zolgensma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Onasemnogene Abeparvovec-xioi (Experimental): Participants will receive a single dose of onasemnogene abeparvovec-xioi, administered intravenously.
  Interventions: Biological: Onasemnogene Abeparvovec-xioi

INTERVENTIONS:
Biological: Onasemnogene Abeparvovec-xioi — Onasemnogene abeparvovec-xioi is a non-replicating recombinant adeno-associated virus serotype 9 (AAV9) containing the human survival motor neuron (SMN) gene under the control of the cytomegalovirus (CMV) enhancer/chicken β-actin-hybrid promoter (CB). Onasemnogene abeparvovec-xioi will be administered as a one-time intravenous infusion over approximately 60 minutes. Dosage will be determined by the participants weight.
  Other Names: Zolgensma

SUMMARY:
This is a Phase 3, open-label, single-arm, single-dose, trial of onasemnogene abeparvovec-xioi (gene replacement therapy) in participants with spinal muscular atrophy (SMA) Type 1 and who are genetically defined by a biallelic pathogenic mutation of the survival motor neuron 1 gene (SMN1) with one or two copies of survival motor neuron 2 gene (SMN2). The primary objective of the study is to evaluate the efficacy of onasemnogene abeparvovec-xioi by assessing the proportion of symptomatic SMA Type 1 participants who achieve the ability to sit unaided for at least 10 seconds up to and including the 18 months of age trial visit. At least 6 participants aged < 6 months (< 180 days) at the time of gene replacement therapy (Day 1) will be enrolled.

DETAILED DESCRIPTION:
This is a Phase 3, open-label, single-arm, single-dose trial of onasemnogene abeparvovec-xioi (gene replacement therapy) in participants with SMA Type 1 with one or 2 copies of SMN2. At least 6 participants < 6 months (< 180 days) of age at the time of gene replacement therapy (Day 1) will be enrolled.

The trial includes 3 trial periods: screening, gene replacement therapy, and follow-up. During the screening period (Days -30 to -2), participants whose parent(s)/legal guardian(s) provide informed consent will undergo screening procedures to determine eligibility for trial enrollment. participants who meet the entry criteria will enter the in-patient gene replacement therapy period (Day -1 to Day 3). On Day -1, participants will be admitted to the hospital for pre-treatment baseline procedures. On Day 1, participants will receive a one-time intravenous (IV) infusion of the equivalent of onasemnogene abeparvovec-xioi cohort 2 dose received in the AVXS-101-CL-101 trial over approximately 60 minutes and will undergo in-patient safety monitoring over the next 48 hours. Participants may be discharged 48 hours after gene replacement therapy, based on Investigator judgment. During the outpatient follow-up period (Days 4 to End of Trial at 18 months of age), participants will return at regularly scheduled intervals for efficacy and safety assessments until the participant reaches 18 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Participants with SMA Type 1 as determined by diagnosis of SMA based on gene mutation analysis with biallelic SMN1 mutations (deletion or point mutations) and one or 2 copies of SMN2 [inclusive of the known SMN2 gene modifier mutation (c.859G>C)]
* Participants must be < 6 months (< 180 days) of age at the time of onasemnogene abeparvovec-xioi infusion
* Participants must have a swallowing evaluation test performed prior to administration of gene replacement therapy
* Up-to-date on childhood vaccinations as per local health authorities.
* Parent(s)/legal guardian(s) willing and able to complete the informed consent process and comply with trial procedures and visit schedule

Exclusion Criteria:

* Previous, planned or expected scoliosis repair surgery/procedure prior to 18 months of age
* Use of invasive ventilatory support (tracheotomy with positive pressure) or pulse oximetry < 95% saturation at screening:

  1. Pulse oximetry saturation must not decrease ≥ 4 percentage points between screening and dosing with confirmatory oximetry reading
  2. Participants may be put on non-invasive ventilatory support for less than 12 hours per day at the discretion of their physician or trial staff
* Use or requirement of non-invasive ventilatory support for greater than or equal to 12 hours daily in the two weeks prior to dosing
* Participant with signs of aspiration based on a swallowing test or whose weight-for-age falls below the 3rd percentile based on World Health Organization (WHO) Child Growth Standards and unwilling to use an alternative method to oral feeding
* Active viral infection (includes human immunodeficiency virus [HIV] or positive serology for hepatitis B, C, or E, or known Zika virus infection)
* Serious non-respiratory tract illness requiring systemic treatment and/or hospitalization within 2 weeks prior to screening
* Upper or lower respiratory infection requiring medical attention, medical intervention, or increase in supportive care of any manner within 4 weeks prior to screening
* Severe non-pulmonary/respiratory tract infection (eg, pyelonephritis, or meningitis) within 4 weeks before administration of gene replacement therapy or concomitant illness that, in the opinion of the Principal Investigator, creates unnecessary risks for gene replacement such as:

  1. Major renal or hepatic impairment
  2. Known seizure disorder
  3. Diabetes mellitus
  4. Idiopathic hypocalcuria
  5. Symptomatic cardiomyopathy
* Known allergy or hypersensitivity to prednisolone or other glucocorticosteroids or their excipients, or human, animal biological raw materials (human transferrin, human insulin, trypsin derived from porcine spleen, bovine derived protein (FBS, bovine milk-derived Benzonase, casamino acid, bovine pancreas), HEK 293 cells, Cosmic Calf Serum, HyQtase) used in manufacturing of onasemnogene abeparvovec-xioi product
* Concomitant use of any of the following: drugs for treatment of myopathy or neuropathy, agents used to treat diabetes mellitus, or ongoing immunosuppressive therapy, plasmapheresis, immunomodulators such as adalimumab, or immunosuppressive therapy within 3 months prior to gene replacement therapy (e.g., corticosteroids, cyclosporine, tacrolimus, methotrexate, cyclophosphamide, IV immunoglobulin, rituximab)
* Anti-AAV9 antibody titer > 1:50 as determined by Enzyme-linked Immunosorbent Assay (ELISA) binding immunoassay. Should a potential participant demonstrate Anti-AAV9 antibody titer > 1:50, he or she may receive retesting within 30 days of the screening period and will be eligible to participate if the Anti-AAV9 antibody titer upon retesting is ≤ 1:50
* Clinically significant abnormal laboratory values (gamma-glutamyl transpeptidase [GGT], ALT, AST, total bilirubin > 2x the ULN, creatinine ≥ 1.0 mg/dL, hemoglobin [Hgb] < 8 or > 18 g/dL; white blood cell [WBC] > 20,000 per cmm) prior to gene replacement therapy. Patients with an elevated bilirubin level that is unequivocally the result of neonatal jaundice shall not be excluded
* Participation in recent SMA treatment clinical trial (with the exception of observational cohort studies or non-interventional studies) or receipt of an investigational or commercial compound, product or therapy administered with the intent to treat SMA (e.g., nusinersen, valproic acid) at any time prior to screening for this trial. Oral beta-agonists must be discontinued at least 30 days prior to dosing. Inhaled albuterol specifically prescribed for the purposes of respiratory (bronchodilator) management is acceptable and not a contraindication at any time prior to screening for this trial
* Expectation of major surgical procedures during the trial assessment period (e.g., spinal surgery or tracheostomy)
* Parent(s)/legal guardian(s) unable or unwilling to comply with trial procedures or inability to travel for repeat visits
* Parent(s)/legal guardian(s) unwilling to keep trial results/observations confidential or to refrain from posting confidential trial results/observations on social media sites
* Parent(s)/legal guardian(s) refuses to sign consent form
* Participants < 35 weeks gestational age at time of birth

Ages: 0 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Tokyo Women's Medical University, Tokyo, Japan
- South Korea (2):
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Seoul National University Hospital, Seoul
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.
URL: https://www.clinicalstudydatarequest.com/.

REFERENCES:
- [Derived] Day JW, Mendell JR, Mercuri E, Finkel RS, Strauss KA, Kleyn A, Tauscher-Wisniewski S, Tukov FF, Reyna SP, Chand DH. Clinical Trial and Postmarketing Safety of Onasemnogene Abeparvovec Therapy. Drug Saf. 2021 Oct;44(10):1109-1119. doi: 10.1007/s40264-021-01107-6. Epub 2021 Aug 12. PMID 34383289
- See also: Novartis Clinical Trial Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17903
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1117

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2 participants took part in the trial at a single site in Taiwan between May 2019 and June 2021.
Pre-assignment Details: A total of 5 participants were screened, of which 3 were screen failures and 2 were enrolled and received study drug.
Groups:
- AVXS-101: Participants received a single dose of AVXS-101 administered as an intravenous (IV) infusion over 60 minutes at a dose of 1.1 × 10^14 vg/kg (vector genome per kilogram) on Day 1 of the overall study. Participants also received daily doses of prophylactic oral prednisolone starting at a dose of 1-2 mg/kg/day from 1 day prior to AVXS-101 infusion until at least 30 days post-infusion at which point the prednisolone dose could be tapered downwards. At week 9, prednisolone could be discontinued.
Period: Overall Study
Arm/Group | AVXS-101
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AVXS-101
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
SMN2 gene modifier mutation (c.859G>C) Present [Count of Participants; unit: Participants] | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Sitting Alone for at Least 10 Seconds
Description: Independent sitting is defined by the World Health Organization Multicentre Growth Reference Study, confirmed by video recording, as a participant who sits up straight unsupported for at least 10 seconds.
Time Frame: From Baseline up to 18 Months of Age Visit
Population: Intent-to-Treat (ITT) population - Symptomatic participants with biallelic deletion mutations of survival of motor neuron 1 (SMN1) (exon 7/8 common homozygous deletions) and 2 copies of survival of motor neuron 2 (SMN2) without the known gene modifier mutation (c.859G>C) who received an IV infusion of AVXS-101 at less than 180 days of age.
Measure: Count of Participants; unit: Participants
Arm/Group | AVXS-101
Number analyzed (Participants) | 2
Participants | 1

2. Secondary Outcome: Event-free Survival at 14 Months of Age
Description: Event-free survival at 14 months of age was defined as the number of participants who did not die, did not require permanent ventilation and did not withdraw from the study by 14 months of age.
Time Frame: From Baseline up to 14 Months of Age
Population: ITT population - Symptomatic participants with biallelic deletion mutations of SMN1 (exon 7/8 common homozygous deletions) and 2 copies of SMN2 without the known gene modifier mutation (c.859G>C) who received an IV infusion of AVXS-101 at less than 180 days of age.
Measure: Count of Participants; unit: Participants
Arm/Group | AVXS-101
Number analyzed (Participants) | 2
Participants | 2

ADVERSE EVENTS:
Time Frame: From Day 1 up to 18 Months of Age Visit (total duration of approximately 12-18 months depending on age at dosing).
Arm/Group | AVXS-101
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AVXS-101 (N=2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AVXS-101 (N=2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (3)
Dysphagia (Gastrointestinal disorders) | 2 (3)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Glucose urine present (Investigations) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1)
Glycosuria (Renal and urinary disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (4)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1)
Urinary tract infection/ (Infections and infestations) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Cleft Palate (Congenital, familial and genetic disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Depending on local requirements, Sponsor's consent necessary before publication of study, or Sponsor can review results communications before public release with a right to request changes to communications regarding trial results between 40 to 60 and up to 90 or 120 days, as applicable, from the time submitted to Sponsor for review to remove references to Sponsor's Confidential Information or delay results communications to permit Sponsor to obtain appropriate Intellectual Property protection.

DOCUMENTS (2):
  • Study Protocol (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT03837184/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/84/NCT03837184/SAP_001.pdf